CLINICAL TRIAL: NCT02629614
Title: Multicenter Study of Safety and Effectiveness of Cala ONE Device for Essential Tremor
Brief Title: Cala ONE Device for Essential Tremor
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cala Health, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ET-03
Record Dates: First submitted 2015-12-08; First posted 2015-12-14 (Estimated); Results first posted 2023-07-18 (Actual); Last update posted 2023-07-18 (Actual); Status verified 2023-06

CONDITIONS: Essential Tremor
MeSH Terms: conditions — Essential Tremor

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- TAPS Stimulation (Experimental): Temporal Afferent Patterned Stimulation (TAPS) is alternating bursts of TENS stimulation applied to the radial and median nerves of a subject's wrist using the Cala ONE device.
  Interventions: Device: Cala ONE Device
- Sham Stimulation (Sham Comparator): 0 amplitude stimulation applied to the radial and median nerves of a subject's wrist using the Cala ONE device.
  Interventions: Device: Cala ONE Device

INTERVENTIONS:
Device: Cala ONE Device — The Cala ONE device is a wrist-worn stimulator which applies transcutaneous electrical stimulation non-invasively to the median and radial nerves of an individual through disposable hydrogel electrodes.

SUMMARY:
This study evaluates the safety and effectiveness of the Cala ONE device to aid in the symptomatic relief of hand tremors in adult essential tremor subjects. This study is a prospective, randomized, double-blinded, sham-controlled study.

ELIGIBILITY:
Inclusion Criteria:

1. 22 years or older
2. A diagnosis of essential tremor as confirmed from clinical history and examination by a movement disorder neurologist
3. Signed informed consent
4. At least one hand exhibiting kinetic tremor ≥ 2 as assessed by the TETRAS Archimedes spiral task completed during the baseline evaluation, as assessed by the Investigator in-person.
5. Score of 3 or above in any one of the items of the Bain & Findley ADL Scale

Exclusion Criteria:

1. Implanted electrical medical device, such as a pacemaker, defibrillator, or deep brain stimulator
2. Previous thalamotomy procedure, including Stereotactic Thalamotomy, Gamma Knife Radiosurgical Thalamotomy, and focused ultrasound, for the treatment of tremor
3. Suspected or diagnosed epilepsy or other seizure disorder
4. Pregnant
5. Swollen, infected, inflamed areas, or skin eruptions, open wounds, or cancerous lesions of skin at stimulation site
6. Peripheral neuropathy affecting the tested upper extremity
7. Alcoholism (score of 4 or higher on DSM-5)
8. Other possible causes of tremor, including Parkinson's disease, drug-induced, enhanced physiological tremor, dystonia
9. Other neurodegenerative disease like Parkinson-plus syndromes suspected on neurological examination. These include: multisystem atrophy, progressive supranuclear palsy, dementia with Lewy bodies, and cortical basal ganglionic degeneration
10. Changes in medication for tremor within 1 month prior to study enrollment
11. Change in antidepressant medication within 3 months prior to study enrollment
12. Botulinum Toxin injection for hand tremor within 6 months prior to study enrollment
13. Current participation in any other interventional research study
14. Previous participation in any other Cala Health interventional research study
15. Alcohol or caffeine consumption within 12 hours of study enrollment

Subjects already taking medications for their essential tremor will remain on their medications during the study with no changes in medication type or dosage levels.

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 93 (Actual)
Dates: Start 2016-04; Primary Completion 2016-11 (Actual); Study Completion 2016-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lin, MD, Study Chair — Clinical Advisor
Locations (4):
- United States (4):
  - UCSF, San Francisco, California
  - The Parkinson's Institute, Sunnyvale, California
  - Kansas University Medical Center, Kansas City, Kansas
  - Swedish Medical Center Seattle, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No
Data will be published, but no PHI will be made available.

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | TAPS Stimulation | Sham Stimulation
Started | 48 | 45
Completed | 48 | 44
Not Completed | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | TAPS Stimulation | Sham Stimulation | Total
Number analyzed (Participants) | 48 | 45 | 93
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 12 | 12 | 24
  >=65 years | 36 | 33 | 69
Age, Continuous [Mean (Standard Deviation); unit: years] | 70.5 (11.2) | 69.8 (10.1) | 70.2 (10.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25 | 23 | 48
  Male | 23 | 22 | 45
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 0 | 2
  Not Hispanic or Latino | 45 | 45 | 90
  Unknown or Not Reported | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 47 | 41 | 88
  More than one race | 1 | 2 | 3
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Change in TETRAS Spiral Rating After Stimulation
Description: The primary effectiveness variable is the change in tremor severity immediately after the stimulation session compared to baseline (immediately prior to stimulation) as measured using the TETRAS Archimedes spiral task (assessed by 3 blinded raters).
  The Essential Tremor Rating Assessment Scale (TETRAS) is a commonly used scale to assess and measure the severity of essential tremor. Each task was calculated individually on a 0-4 scale, with higher scores indicating more severe tremors.
Time Frame: Immediately before and after 40 minute stimulation session
Population: Of the 92 subjects that completed the study, 77 were included in the analysis. 15 (8 in the treatment group and 7 in the sham group) were excluded due to significant protocol deviation reasons.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | TAPS Stimulation | Sham Stimulation
Number analyzed (Participants) | 40 | 37
score on a scale
  Baseline | 2.95 (0.68) | 2.63 (0.52)
  Post Stimulation | 2.41 (1) | 2.23 (0.80)

2. Secondary Outcome: Change in TETRAS Spiral Rating During Stimulation
Description: An additional analysis variable is the change in tremor severity during the stimulation session (30 minutes into stimulation session) compared to baseline (immediately prior to stimulation) as measured using the TETRAS Archimedes spiral task (assessed by 3 blinded raters).
  The Essential Tremor Rating Assessment Scale (TETRAS) is a commonly used scale to assess and measure the severity of essential tremor. Each task was calculated individually on a 0-4 scale, with higher scores indicating more severe tremors.
Time Frame: Immediately before and 30 minutes into stimulation session
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | TAPS Stimulation | Sham Stimulation
Number analyzed (Participants) | 40 | 37
score on a scale
  Baseline | 2.95 (0.68) | 2.63 (0.52)
  During Stimulation | 2.58 (0.90) | 2.26 (0.67)

3. Secondary Outcome: Self-report Improvement
Description: The percentage of subjects in the treatment group indicating improvement on the CGI-I Scale will be compared to the sham group. The Clinical Global Impression - Improvement (GGI-I) scale evaluates a clinician's rating of tremor improvement noted in the subject, as a result of the treatment. The scale ranges from 1 (very much improved) to 7 (very much worse).
Time Frame: Immediately before and after 40 minute stimulation session
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | TAPS Stimulation | Sham Stimulation
Number analyzed (Participants) | 40 | 37
Participants | 35 | 23

4. Other Pre Specified Outcome: Change in Kinetic Tremor
Description: The change in tremor severity on the kinetic tremor task as assessed by an investigator using the TETRAS rating scale.
  The Essential Tremor Rating Assessment Scale (TETRAS) is a commonly used scale to assess and measure the severity of essential tremor. Each task was calculated individually on a 0-4 scale, with higher scores indicating more severe tremors.
Time Frame: Immediately before and after 40 minute stimulation session
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | TAPS Stimulation | Sham Stimulation
Number analyzed (Participants) | 40 | 37
score on a scale
  Baseline | 2.29 (0.47) | 2.27 (0.47)
  Change after stimulation | -0.53 (0.59) | -0.34 (0.43)

5. Other Pre Specified Outcome: Change in Kinetic Tremor
Description: as for outcome 4
Time Frame: Immediately before and 30 minutes into stimulation session
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | TAPS Stimulation | Sham Stimulation
Number analyzed (Participants) | 40 | 37
score on a scale
  Baseline | 2.29 (0.47) | 2.27 (0.47)
  Change during stimulation | -0.50 (0.51) | -0.53 (0.59)

6. Other Pre Specified Outcome: Change in Lateral "Wing Beating" Postural Tremor
Description: The change in tremor severity in the lateral "wing beating" postural tremor task as assessed by an investigator using the TETRAS rating scale.
  The Essential Tremor Rating Assessment Scale (TETRAS) is a commonly used scale to assess and measure the severity of essential tremor. Each task was calculated individually on a 0-4 scale, with higher scores indicating more severe tremors.
Time Frame: Immediately before and after 40 minute stimulation session
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | TAPS Stimulation | Sham Stimulation
Number analyzed (Participants) | 40 | 37
score on a scale
  Baseline | 2.29 (0.70) | 2.16 (0.57)
  Change after stimulation | -0.56 (0.72) | -0.36 (0.54)

7. Other Pre Specified Outcome: Change in Lateral "Wing Beating" Postural Tremor
Description: as for outcome 6
Time Frame: Immediately before and 30 minutes into stimulation session
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | TAPS Stimulation | Sham Stimulation
Number analyzed (Participants) | 40 | 37
score on a scale
  Baseline | 2.29 (0.70) | 2.16 (0.57)
  Change during stimulation | -0.51 (0.70) | -0.34 (0.44)

8. Other Pre Specified Outcome: Change in Forward Outstretched Postural Tremor
Description: The change in tremor severity on outstretched tremor task as assessed by an investigator using the TETRAS rating scale.
  The Essential Tremor Rating Assessment Scale (TETRAS) is a commonly used scale to assess and measure the severity of essential tremor. Each task was calculated individually on a 0-4 scale, with higher scores indicating more severe tremors.
Time Frame: Immediately before and after 40 minute stimulation session
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | TAPS Stimulation | Sham Stimulation
Number analyzed (Participants) | 40 | 37
score on a scale
  Baseline | 1.96 (0.54) | 1.91 (0.54)
  Change after stimulation | -0.75 (0.65) | -0.35 (0.51)

9. Other Pre Specified Outcome: Change in Forward Outstretched Postural Tremor
Description: as for outcome 8
Time Frame: Immediately before and 30 minutes into stimulation session
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | TAPS Stimulation | Sham Stimulation
Number analyzed (Participants) | 40 | 37
score on a scale
  Baseline | 1.96 (0.54) | 1.91 (0.54)
  Change during stimulation | -0.56 (0.59) | -0.35 (0.41)

10. Other Pre Specified Outcome: Change in Bain & Findley ADL: Use a Spoon to Drink Liquid
Description: The change in tremor severity on drinking liquid with a spoon as assessed by the subject using the Bain & Findley ADL rating scale.
  The Bain and Findley Activities of Daily Living (BF-ADL) assessment evaluates the subject's ability to perform a number of specific ADLs, measured before and after treatment. Each ADL is performed by the subject and self-rated on a scale of 1-4, with higher scores indicating greater difficulty in performing the task.
Time Frame: Immediately before and after 40 minute stimulation session
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | TAPS Stimulation | Sham Stimulation
Number analyzed (Participants) | 40 | 37
score on a scale
  Baseline | 3.18 (0.78) | 3.00 (0.85)
  Change after stimulation | -0.78 (0.89) | -0.59 (0.76)

11. Other Pre Specified Outcome: Change in Bain & Findley ADL: Hold a Cup of Liquid
Description: The change in tremor severity on holding a cup of liquid as assessed by the subject using the Bain & Findley ADL rating scale.
  The Bain and Findley Activities of Daily Living (BF-ADL) assessment evaluates the subject's ability to perform a number of specific ADLs, measured before and after treatment. Each ADL is performed by the subject and self-rated on a scale of 1-4, with higher scores indicating greater difficulty in performing the task.
Time Frame: Immediately before and after 40 minute stimulation session
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | TAPS Stimulation | Sham Stimulation
Number analyzed (Participants) | 40 | 37
score on a scale
  Baseline | 2.95 (0.85) | 2.65 (0.92)
  Change after stimulation | -1.03 (0.73) | -0.57 (0.80)

12. Other Pre Specified Outcome: Change in Bain & Findley ADL: Pouring
Description: The change in tremor severity on pouring as assessed by the subject using the Bain & Findley ADL rating scale.
  The Bain and Findley Activities of Daily Living (BF-ADL) assessment evaluates the subject's ability to perform a number of specific ADLs, measured before and after treatment. Each ADL is performed by the subject and self-rated on a scale of 1-4, with higher scores indicating greater difficulty in performing the task.
Time Frame: Immediately before and after 40 minute stimulation session
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | TAPS Stimulation | Sham Stimulation
Number analyzed (Participants) | 40 | 37
score on a scale
  Baseline | 2.78 (1.03) | 2.59 (0.86)
  Change after stimulation | -0.70 (0.76) | -0.59 (0.72)

13. Other Pre Specified Outcome: Change in Bain & Findley ADL: Dialing
Description: The change in tremor severity on dialing a telephone as assessed by the subject using the Bain & Findley ADL rating scale.
  The Bain and Findley Activities of Daily Living (BF-ADL) assessment evaluates the subject's ability to perform a number of specific ADLs, measured before and after treatment. Each ADL is performed by the subject and self-rated on a scale of 1-4, with higher scores indicating greater difficulty in performing the task.
Time Frame: Immediately before and after 40 minute stimulation session
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | TAPS Stimulation | Sham Stimulation
Number analyzed (Participants) | 40 | 37
score on a scale
  Baseline | 2.23 (0.89) | 2.00 (0.91)
  Change after stimulation | -0.70 (0.79) | -0.30 (0.62)

14. Other Pre Specified Outcome: Change in Bain & Findley ADL: Picking up Change
Description: The change in tremor severity on picking up change as assessed by the subject using the Bain & Findley ADL rating scale.
  The Bain and Findley Activities of Daily Living (BF-ADL) assessment evaluates the subject's ability to perform a number of specific ADLs, measured before and after treatment. Each ADL is performed by the subject and self-rated on a scale of 1-4, with higher scores indicating greater difficulty in performing the task.
Time Frame: Immediately before and after 40 minute stimulation session
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | TAPS Stimulation | Sham Stimulation
Number analyzed (Participants) | 40 | 37
score on a scale
  Baseline | 2.03 (0.86) | 1.92 (0.89)
  Change after stimulation | -0.53 (0.68) | -0.05 (0.62)

15. Other Pre Specified Outcome: Change in Bain & Findley ADL: Inserting Plug Into Socket
Description: The change in tremor severity on inserting a plug into a socket as assessed by the subject using the Bain & Findley ADL rating scale.
  The Bain and Findley Activities of Daily Living (BF-ADL) assessment evaluates the subject's ability to perform a number of specific ADLs, measured before and after treatment. Each ADL is performed by the subject and self-rated on a scale of 1-4, with higher scores indicating greater difficulty in performing the task.
Time Frame: Immediately before and after 40 minute stimulation session
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | TAPS Stimulation | Sham Stimulation
Number analyzed (Participants) | 40 | 37
score on a scale
  Baseline | 1.83 (0.78) | 1.76 (0.80)
  Change after stimulation | -0.33 (0.69) | -0.24 (0.55)

16. Other Pre Specified Outcome: Change in Bain & Findley ADL: Unlocking
Description: The change in tremor severity on unlocking a lock with a key as assessed by the subject using the Bain & Findley ADL rating scale.
  The Bain and Findley Activities of Daily Living (BF-ADL) assessment evaluates the subject's ability to perform a number of specific ADLs, measured before and after treatment. Each ADL is performed by the subject and self-rated on a scale of 1-4, with higher scores indicating greater difficulty in performing the task.
Time Frame: Immediately before and after 40 minute stimulation session
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | TAPS Stimulation | Sham Stimulation
Number analyzed (Participants) | 40 | 37
score on a scale
  Baseline | 2.23 (0.86) | 1.86 (0.67)
  Change after stimulation | -0.60 (0.87) | -0.16 (0.55)

ADVERSE EVENTS:
Arm/Group | TAPS Stimulation | Sham Stimulation
Serious Adverse Events (participants affected / at risk) | 0/48 | 0/45
Other Adverse Events (participants affected / at risk) | 2/48 | 1/45
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | TAPS Stimulation (N=48) | Sham Stimulation (N=45)
Skin Irritation (Skin and subcutaneous tissue disorders) | 2 | 0
Feeling of weakness around the wrist (Nervous system disorders) | 1 | 0
Stinging pain in wrist (Skin and subcutaneous tissue disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No